CLINICAL TRIAL: NCT02102776
Title: Intraoperative Mitomycin C Application, Amniotic Membrane Transplantation and Conjunctival Autograft After Primary Pterygium Excision: A Multi-center Randomized Clinical Trial
Brief Title: Intraoperative Mitomycin C, Amniotic Membrane Transplantation and Conjunctival Autograft for Primary Pterygium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shiyou Zhou, M.D., Ph.D, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014015
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Pterygium
Keywords: Primary Pterygium; Mitomycin C; Amniotic membrane transplantation; Conjunctival autograft; Multi-center randomized clinical trial
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MMC after pterygium excision (Active Comparator): Intraoperative mitomycin C (0.02%) will be applied for 5 minutes after pterygium excision. The conjunctival defect will be left bare without graft.
  Interventions: Procedure: MMC; Procedure: Pterygium excision
- AMT after Pterygium Excision (Active Comparator): Amniotic membrane transplantation will be applied to cover the conjunctival defect after pterygium excision. No mitomycin C will be applied.
  Interventions: Procedure: AMT; Procedure: Pterygium excision
- CAG after Pterygium Excision (Active Comparator): A conjunctival autograft will be harvested from the superior side of the operating eye's bulbar conjunctiva. Then the graft will be sutured to cover the conjunctival defect after pterygium excision. No mitomycin C will be applied.
  Interventions: Procedure: CAG; Procedure: Pterygium excision

INTERVENTIONS:
Procedure: MMC — Standardized cotton soaked in mitomycin C (0.02%) will be applied underneath conjunctiva for 5 minutes after pterygium excision.
  Other Names: Intraoperative mitomycin C
  Arms: MMC after pterygium excision
Procedure: AMT — Amniotic membrane transplantation will be applied to cover the conjunctival defect after pterygium excision.
  Other Names: Amniotic membrane transplantation
  Arms: AMT after Pterygium Excision
Procedure: CAG — A conjunctival autograft, harvested from the superior bulbar conjunctiva of the operating eye, will be applied to cover the conjunctival defect after pterygium excision.
  Other Names: Conjunctival autograft
  Arms: CAG after Pterygium Excision
Procedure: Pterygium excision — Pterygium head, minimal conjunctiva and anterior tenon's capsule underneath will be removed in the excision of pterygium tissue.

SUMMARY:
The purpose of this randomized multi-center clinical trial is to compare the efficacy and safety of intraoperative mitomycin C(MMC),amniotic membrane transplantation(AMT) and Conjunctival Autograft(CAG) for primary pterygium surgery. The investigators will also evaluate particular risk factors related to pterygium recurrence.

DETAILED DESCRIPTION:
Patients with primary pterygium will be randomly assigned to undertake pterygium excision followed by intraoperative mitomycin C application,amniotic membrane transplantation or conjunctival autograft in five clinical centers. Multi-center collaboration and quality monitoring will be based on a website designed for this study. The patients will be followed at least 12 months. Corneal Recurrence as the primary outcome measure, is considered as a fibrovascular ingrowth beyond the limbus with conjunctival drag.

ELIGIBILITY:
Inclusion Criteria:

* Primary pterygium
* Willingness to participate in research project and to attend research follow-up
* Adults (age 18 to 80 years old)
* Patients must not meet any of the following exclusion criteria

Exclusion Criteria:

* Pregnant,breast-feeding women or patients with poor general health
* Patients with significant ocular or lid pathology, such as Sjogren's Syndrome, infection, exposure keratitis, glaucoma, active uveitis, retinal detachment and trauma
* Patients with previous surgery on ocular surface, such as trabeculectomy, strabismus surgery
* Patients with allergy to intraoperative or postoperative drugs, such as mitomycin C, tobramycin or local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pterygium | One year
  Corneal Recurrence is considered as a fibrovascular ingrowth beyond the limbus with conjunctival drag

SECONDARY OUTCOMES:
Visual acuity | One year
Healing time of corneal epithelium | Four weeks
Healing time of conjunctival epithelium | Four weeks
Postoperative complications | One year

CONTACTS AND LOCATIONS:
Overall Officials: Shiyou Zhou, M.D., Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (5):
- China (5):
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xi'an Eye Hospital, Xi’an, Shanxi
  - Sichuan Ganzi Autonomous Prefecture People's Hospital, Ganzi, Sichuan
  - The Fourth Affiliated Hospital, Kunming Medical University, Kunming, Yunnan